CLINICAL TRIAL: NCT04014361
Title: Single- and Multiple-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study With LY3154885 in Healthy Subjects
Brief Title: A Study of LY3154885 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: HUAA study is terminated early due to a business decision.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17051; J1Z-MC-HUAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- LY3154885 - Part A (Experimental): 15, 45, 100, 200, 300 or 375 milligrams (mg) LY3154885 administered orally in two of three study periods.
  Interventions: Drug: LY3154885 - Capsule
- Placebo - Part A (Placebo Comparator): Placebo administered orally in one of three study periods.
  Interventions: Drug: Placebo - Capsule
- 45 mg LY3154885 + Itraconazole - Part B (Experimental): 45 mg LY3154885 administered orally in period 1 followed by 200 mg Itraconazole administered orally on 10 consecutive days and then 45 mg LY3154885 co-administered with 200 mg itraconazole orally during period 2.
  Interventions: Drug: LY3154885 - Capsule; Drug: Itraconazole
- Placebo + Itraconazole - Part B (Placebo Comparator): Placebo administered orally during period 1 followed by 200 mg Itraconazole administered orally on 10 consecutive days and then placebo co-administered with 200 mg itraconazole orally during period 2.
  Interventions: Drug: Placebo - Capsule; Drug: Itraconazole
- LY3154885 - Part C (Experimental): Part C was not initiated.
  Interventions: Drug: LY3154885 - Capsule
- Placebo - Part C (Placebo Comparator): Part C was not initiated.
  Interventions: Drug: Placebo - Capsule
- LY3154885 - Part D (Experimental): Part D was not initiated.
  Interventions: Drug: LY3154885 - Capsule; Drug: LY3154885 - Tablet

INTERVENTIONS:
Drug: LY3154885 - Capsule — Administered orally.
  Arms: 45 mg LY3154885 + Itraconazole - Part B; LY3154885 - Part A; LY3154885 - Part C; LY3154885 - Part D
Drug: Placebo - Capsule — Administered orally.
  Arms: Placebo + Itraconazole - Part B; Placebo - Part A; Placebo - Part C
Drug: Itraconazole — Administered orally.
  Arms: 45 mg LY3154885 + Itraconazole - Part B; Placebo + Itraconazole - Part B
Drug: LY3154885 - Tablet — Administered orally.
  Arms: LY3154885 - Part D

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of LY3154885 when given by mouth to healthy participants. The study will have up to four parts. Each participant will enroll in only one part. The study will last up to 70 days for each participant, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Male participants:

  * Men, regardless of their fertility status, with partners who are nonpregnant women of childbearing potential, must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use condoms with spermicide as well as 1 additional highly effective (<1% failure rate) method of contraception or effective method of contraception (such as diaphragms with spermicide) for 3 months following dosing
  * Men with pregnant partners should use condoms with spermicide during intercourse for the duration of the study or for 3 months following dosing, whichever is longer
  * Men who are in exclusively same-sex relationships (as their preferred and usual lifestyle) or with female partners of non-childbearing potential are not required to use contraception
  * Men should refrain from sperm donation for the duration of the study or for 3 months following the last dose of study drug, whichever is longer
* Female participants of non-childbearing potential, including those who are:

  * Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, confirmed tubal ligation, or tubal occlusion) or congenital anomaly such as Müllerian agenesis; or
  * Postmenopausal, defined as 1 of the following:

    * A woman at least 50 years of age with an intact uterus, not on hormone replacement therapy, who has had either:

      * Cessation of menses for at least 1 year; or
      * At least 6 months of spontaneous amenorrhea with a follicle-stimulating hormone level ≥40 milli-international units per milliliter (mIU/mL) at screening
    * A woman at least 55 years of age, not on hormone replacement therapy, who has had at least 6 months of spontaneous amenorrhea; or
    * A woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy
* Have a body mass index (BMI) of 18.0 to 35.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Have a marked baseline prolongation of/corrected QT (QTc) interval (for example, repeated demonstration of a QTcB interval >450 milliseconds [msec] for males or >470 msec for females);

  * A history of additional risk factors for Torsades de Pointes (for example, heart failure, hypokalemia, family history of Long QT Syndrome);
  * The use of concomitant medications that prolong the QT/QTc interval
* Have an abnormal blood pressure (BP) (taken after the participant has been in a supine position for at least 5 minutes) for the population, as determined by a systolic BP >140 millimeters of mercury (mmHg) or a diastolic BP >90 mmHg at screening or a preexisting history of hypertension. Up to 2 additional measurements may be taken after an appropriate resting interval at screening to confirm eligibility
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (such as Cushing syndrome, hyperthyroidism, hyperaldosteronism), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational medicinal product (IMP); or of interfering with the interpretation of data
* Have a history of or current significant psychiatric disorders

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885): Period 1:
  Participants received Placebo administered orally on Day 1.
  Period 2:
  Participants received 100 milligrams (mg) LY3154885 administered orally on Day 1.
  Period 3:
  Participants received 375 mg LY3154885 administered orally on Day 1.
- Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885): Period 1:
  Participants received 15 mg LY3154885 administered orally on Day 1.
  Period 2:
  Participants received Placebo administered orally on Day 1
  Period 3:
  Participants received 375 mg LY3154885 administered orally on Day 1.
- Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo): Period 1:
  Participants received 15 mg LY3154885 administered orally on Day 1.
  Period 2:
  Participants received 100 mg LY3154885 administered orally on Day 1.
  Period 3:
  Participants received Placebo administered orally on Day 1.
- Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo): Period 1:
  Participants received 45 mg LY3154885 administered orally on Day 1.
  Period 2:
  Participants received 200 mg LY3154885 administered orally on Day 1.
  Period 3:
  Participants received Placebo administered orally on Day 1.
- Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885): Period 1:
  Participants received Placebo administered orally on Day 1.
  Period 2:
  Participants received 200 mg LY3154885 administered orally on Day 1.
  Period 3:
  Participants received 300 mg LY3154885 administered orally on Day 1.
- Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885): Period 1:
  Participants received 45 mg LY3154885 administered orally on Day 1.
  Period 2:
  Participants received Placebo administered orally on Day 1.
  Period 3:
  Participants received 300 mg LY3154885 administered orally on Day 1
- Part B: 45 LY3154885 + 200 mg Itraconazole: Period 1:
  Participants received 45 mg LY3154885 administered orally.
  Period 2:
  Participants received 200 mg Itraconazole administered orally on 10 consecutive days and then 45 mg LY3154885 co-administered with 200 mg itraconazole orally.
- Part B: Placebo + 200 mg Itraconazole: Period 1:
  Participants received placebo administered orally.
  Period 2:
  Participants received 200 mg Itraconazole administered orally on 10 consecutive days and then placebo co-administered with 200 mg itraconazole orally.
Period: Period 1
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Started | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Received at Least One Dose of Study Drug | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (7 Days)
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Started | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Started | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3
Completed | 4 | 4 | 4 | 3 | 4 | 4 | 9 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout 2 (7 Days)
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Started | 4 | 4 | 4 | 3 | 4 | 4 | 0 (Part B had only two periods.) | 0 (Part B had only two periods.)
Completed | 4 | 4 | 4 | 3 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Started | 4 | 4 | 4 | 3 | 4 | 4 | 0 | 0
Completed | 4 | 4 | 4 | 3 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885): Period 1:
  Participants received Placebo administered orally on Day 1.
  Period 2:
  Participants received 100 mg LY3154885 administered orally on Day 1.
  Period 3:
  Participants received 375 mg LY3154885 administered orally on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1, Sequence 1 (Placebo, 100 mg LY3154885, 375 mg LY3154885) | Part A: Cohort 1, Sequence 2 (15 mg LY3154885, Placebo, 375 mg LY3154885) | Part A: Cohort 1, Sequence 3 (15 mg LY3154885, 100 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 1 (45 mg LY3154885, 200 mg LY3154885, Placebo) | Part A: Cohort 2, Sequence 2 (Placebo, 200 mg LY3154885, 300 mg LY3154885) | Part A: Cohort 2, Sequence 3 (45 mg LY3154885, Placebo, 300 mg LY3154885) | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 9
  Male | 3 | 3 | 3 | 2 | 1 | 3 | 9 | 3 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 0 | 1 | 0 | 2 | 1 | 9
  Not Hispanic or Latino | 3 | 3 | 1 | 4 | 3 | 4 | 7 | 2 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 4 | 2 | 4 | 4 | 1 | 20
  White | 2 | 2 | 3 | 0 | 2 | 0 | 5 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 9 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any AE from this study that results in one of the following: death, initial or prolonged inpatient hospitalization, a life-threatening experience (that is, immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Time Frame: Baseline through Study Completion (Up to 5 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Placebo: Participants received Placebo administered orally.
- Part A 15 mg LY3154885: Participants received 15 mg LY3154885 administered orally.
- Part A 45 mg LY3154885: Participants received 45 mg LY3154885 administered orally.
- Part A 100 mg LY3154885: Participants received 100 mg LY3154885 administered orally.
- Part A 200 mg LY3154885: Participants received 200 mg LY3154885 administered orally.
- Part A 300 mg LY3154885: Participants received 300 mg LY3154885 administered orally.
- Part A 375 mg LY3154885: Participants received 375 mg LY3154885 administered orally.
Arm/Group | Part A Placebo | Part A 15 mg LY3154885 | Part A 45 mg LY3154885 | Part A 100 mg LY3154885 | Part A 200 mg LY3154885 | Part A 300 mg LY3154885 | Part A 375 mg LY3154885 | Part B: 45 LY3154885 + 200 mg Itraconazole | Part B: Placebo + 200 mg Itraconazole
Number analyzed (Participants) | 23 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3154885
Description: Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3154885
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post dose
Population: Part A: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part A 15 mg LY3154885 | Part A 45 mg LY3154885 | Part A 100 mg LY3154885 | Part A 200 mg LY3154885 | Part A 300 mg LY3154885 | Part A 375 mg LY3154885
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 8
Nanograms per milliliter (ng/mL) | 95.7 (35) | 156 (43) | 519 (39) | 763 (69) | 1180 (38) | 1360 (43)

3. Secondary Outcome: Part B: PK: Maximum Concentration (Cmax) of LY3154885
Description: Part B: PK: Maximum Concentration (Cmax) of LY3154885
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post dose; Day 14: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72 and 96 hours post dose.
Population: Part B: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B 45 mg LY3154885: Participants received 45 mg LY3154885 administered orally.
- Part B 45 mg LY3154885 + 200 mg Itraconazole: Participants received 45 mg LY3154885 + 200 mg Itraconazole administered orally.
Arm/Group | Part B 45 mg LY3154885 | Part B 45 mg LY3154885 + 200 mg Itraconazole
Number analyzed (Participants) | 9 | 9
ng/mL
  LY3154885 Single Dose (Day 1) | 219 (52) | NA (NA) — Reporting only LY3154885 Single Dose (Day 1) data on this row
  LY3154885 Single Dose + Itraconazole QD (Day 14) | NA (NA) — Reporting only LY3154885 Single Dose + Itraconazole QD (Day 14) on this row. | 408 (33)

4. Secondary Outcome: Part A, PK: Time to Maximum Plasma Concentration (Tmax) LY3154885
Description: Part A, PK: Time to Maximum Plasma Concentration (Tmax) LY3154885
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post dose
Population: Part A: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A 15 mg LY3154885 | Part A 45 mg LY3154885 | Part A 100 mg LY3154885 | Part A 200 mg LY3154885 | Part A 300 mg LY3154885 | Part A 375 mg LY3154885
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 8
Hours | 3.00 [2.00 to 3.08] | 4.00 [2.00 to 5.00] | 3.01 [2.00 to 5.05] | 3.00 [2.00 to 6.05] | 3.00 [2.00 to 6.00] | 3.02 [2.00 to 5.00]

5. Secondary Outcome: Part B, PK: Time to Maximum Plasma Concentration (Tmax) LY3154885
Time Frame: as for outcome 3
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B 45 mg LY3154885 | Part B 45 mg LY3154885 + 200 mg Itraconazole
Number analyzed (Participants) | 9 | 9
Hours
  LY3154885 Single Dose (Day 1) | 2.00 [1.00 to 8.00] | NA [NA to NA] — Reporting only LY3154885 Single Dose (Day 1) data on this row.
  LY3154885 Single Dose + Itraconazole QD (Day 14) | NA [NA to NA] — Reporting only LY3154885 Single Dose + Itraconazole QD (Day 14) on this row. | 6.00 [3.00 to 8.03]

6. Secondary Outcome: Part A, PK: Area Under the Concentration Versus Time Curve to Infinity [AUC(0-∞)] of LY3154885
Description: Part A, PK: Area Under the Concentration Versus Time Curve to Infinity [AUC(0-∞)] of LY3154885
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 hours post dose
Population: Part A: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (h*ng/mL)
Arm/Group | Part A 15 mg LY3154885 | Part A 45 mg LY3154885 | Part A 100 mg LY3154885 | Part A 200 mg LY3154885 | Part A 300 mg LY3154885 | Part A 375 mg LY3154885
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 8
nanogram hour per milliliter (h*ng/mL) | 1290 (53) | 2710 (48) | 8410 (59) | 14900 (96) | 30900 (82) | 28600 (48)

7. Secondary Outcome: Part B, PK: Area Under the Concentration Versus Time Curve to Infinity [AUC(0-∞)] of LY3154885
Description: Part B, PK: Area Under the Concentration Versus Time Curve to Infinity [AUC(0-∞)] of LY3154885
Time Frame: as for outcome 3
Population: Part B: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part B: 45 mg LY3154885: Participants received 45 mg LY3154885 administered orally.
- Part B: 45 mg LY3154885 + 200 mg Itraconazole: Participants received 45 mg LY3154885 + 200 mg Itraconazole administered orally.
Arm/Group | Part B: 45 mg LY3154885 | Part B: 45 mg LY3154885 + 200 mg Itraconazole
Number analyzed (Participants) | 9 | 9
h*ng/mL
  LY3154885 Single Dose (Day 1) | 4510 (54) | NA (NA) — Reporting only LY3154885 Single Dose (Day 1) data on this row.
  LY3154885 Single Dose + Itraconazole QD (Day 14) | NA (NA) — Reporting only LY3154885 Single Dose + Itraconazole QD (Day 14) on this row | 16900 (34)

ADVERSE EVENTS:
Time Frame: Baseline Up To 5 Months
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Part B Placebo: Participants received Placebo administered orally.
- Part B 200 mg Itraconazole: Participants received 200 mg Itraconazole administered orally.
- Part B Placebo + 200 mg Itraconazole: Participants received Placebo + 200 mg Itraconazole administered orally.
Arm/Group | Part A Placebo | Part A 15 mg LY3154885 | Part A 45 mg LY3154885 | Part A 100 mg LY3154885 | Part A 200 mg LY3154885 | Part A 300 mg LY3154885 | Part A 375 mg LY3154885 | Part B Placebo | Part B 45 mg LY3154885 | Part B 200 mg Itraconazole | Part B 45 mg LY3154885 + 200 mg Itraconazole | Part B Placebo + 200 mg Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/3 | 0/9 | 0/12 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/3 | 0/9 | 0/12 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 2/23 | 0/8 | 0/8 | 1/8 | 0/8 | 2/8 | 6/8 | 0/3 | 0/9 | 1/12 | 1/9 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Placebo (N=23) | Part A 15 mg LY3154885 (N=8) | Part A 45 mg LY3154885 (N=8) | Part A 100 mg LY3154885 (N=8) | Part A 200 mg LY3154885 (N=8) | Part A 300 mg LY3154885 (N=8) | Part A 375 mg LY3154885 (N=8) | Part B Placebo (N=3) | Part B 45 mg LY3154885 (N=9) | Part B 200 mg Itraconazole (N=12) | Part B 45 mg LY3154885 + 200 mg Itraconazole (N=9) | Part B Placebo + 200 mg Itraconazole (N=3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A strategic business decision was made to terminate the study prior to initiation of the multiple-ascending dose study (Part C). The secondary objectives pertaining to Part D were not evaluated as the study was terminated before the commencement of Part D.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT04014361/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT04014361/SAP_001.pdf